CLINICAL TRIAL: NCT01652703
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate Tolerability and Efficacy of AMG 145 on LDL-C in Combination With Stable Statin Therapy in Japanese Subjects With Hypercholesterolemia and High Cardiovascular Risk
Brief Title: A Study to Evaluate Tolerability and Efficacy of Evolocumab (AMG 145) in Japanese Subjects
Acronym: AMG145
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20110231
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Hypercholesterolemia and High Risk for Cardiovascular Events
Keywords: Japanese, hypercholesterolemia, high risk for cardiovascular events
MeSH Terms: conditions — Hypercholesterolemia | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo Q2W (Placebo Comparator): Participants received placebo subcutaneous injection once every 2 weeks (Q2W) for 12 weeks.
  Interventions: Other: Placebo
- Placebo Q4W (Placebo Comparator): Participants received placebo subcutaneous injection once every 4 weeks (Q4W) for 12 weeks.
  Interventions: Other: Placebo
- Evolocumab 70 mg Q2W (Experimental): Participants received 70 mg evolocumab by subcutaneous injection once every 2 weeks for 12 weeks.
  Interventions: Biological: Evolocumab
- Evolocumab 140 mg Q2W (Experimental): Participants received 140 mg evolocumab by subcutaneous injection once every 2 weeks for 12 weeks.
  Interventions: Biological: Evolocumab
- Evolocumab 280 mg Q4W (Experimental): Participants received 280 mg evolocumab by subcutaneous injection once every 4 weeks for 12 weeks.
  Interventions: Biological: Evolocumab
- Evolocumab 420 mg Q4W (Experimental): Participants received 420 mg evolocumab by subcutaneous injection once every 4 weeks for 12 weeks.
  Interventions: Biological: Evolocumab

INTERVENTIONS:
Biological: Evolocumab — Administered by subcutaneous injection
  Other Names: AMG 145; Repatha
  Arms: Evolocumab 140 mg Q2W; Evolocumab 280 mg Q4W; Evolocumab 420 mg Q4W; Evolocumab 70 mg Q2W
Other: Placebo — Administered by subcutaneous injection
  Arms: Placebo Q2W; Placebo Q4W

SUMMARY:
The primary objective is to evaluate the effect of 12 weeks of subcutaneous evolocumab every 2 weeks or every 4 weeks, compared with placebo, on percent change from baseline in low-density lipoprotein cholesterol (LDL-C) when used in addition to statin therapy in Japanese adults with hypercholesterolemia and high cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria: Japanese adult, on statin, with or without ezetimibe, with stable dose(s) for at least 4 weeks, fasting LDL-C greater than or equal to 115 mg/dL (3.0 mmol/L), fasting triglycerides less than or equal to 400 mg/dL (4.5 mmol/L); Exclusion Criteria: New York Heart Association (NYHA) class III or IV, poorly controlled hypertension, recently diagnosed or poorly controlled type 2 diabetes, last known left ventricular ejection fraction < 30%, myocardial infarction, unstable angina, percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG), stroke, planned cardiac surgery or revascularization within 6 months of randomization, uncontrolled cardiac arrhythmia.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2012-07-10 (Actual); Primary Completion 2013-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (35):
- Japan (35):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Fukui-shi, Fukui
  - Research Site, Kasuga-shi, Fukuoka
  - Research Site, Gifu, Gifu
  - Research Site, Fujioka-shi, Gunma
  - Research Site, Maebashi, Gunma
  - Research Site, Takasaki-shi, Gunma
  - Research Site, Kawanishi, Hyōgo
  - Research Site, Kobe, Hyōgo
  - Research Site, Hitachi-shi, Ibaraki
  - Research Site, Koga-shi, Ibaraki
  - Research Site, Mito, Ibaraki
  - Research Site, Komatsu-shi, Ishikawa-ken
  - Research Site, Takamatsu, Kagawa-ken
  - Research Site, Kochi, Kochi
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Kyoto, Kyoto
  - Research Site, Ina-shi, Nagano
  - Research Site, Matsumoto-shi, Nagano
  - Research Site, Suwa-shi, Nagano
  - Research Site, Ibaraki-shi, Osaka
  - Research Site, Suita-shi, Osaka
  - Research Site, Toyonaka-shi, Osaka
  - Research Site, Hanyu-shi, Saitama
  - Research Site, Sayama-shi, Saitama
  - Research Site, Toda-shi, Saitama
  - Research Site, Ōtsu, Shiga
  - Research Site, Bunkyo-ku, Tokyo
  - Research Site, Chiyoda-ku, Tokyo
  - Research Site, Chuo-ku, Tokyo
  - Research Site, Hachioji-shi, Tokyo
  - Research Site, Itabashi-ku, Tokyo
  - Research Site, Shinagawa-ku, Tokyo
  - Research Site, Taito-ku, Tokyo
  - Research Site, Toshima-ku, Tokyo

REFERENCES:
- [Background] Hirayama A, Yamashita S, Inomata H, Kassahun H, Cyrille M, Ruzza A, Yoshida M, Kiyosue A, Ma Y, Teramoto T. One-Year Efficacy and Safety of Evolocumab in Japanese Patients - A Pooled Analysis From the Open-Label Extension OSLER Studies. Circ J. 2017 Jun 23;81(7):1029-1035. doi: 10.1253/circj.CJ-16-1016. Epub 2017 Mar 29. PMID 28367845
- [Background] Toth PP, Descamps O, Genest J, Sattar N, Preiss D, Dent R, Djedjos C, Wu Y, Geller M, Uhart M, Somaratne R, Wasserman SM; PROFICIO Investigators. Pooled Safety Analysis of Evolocumab in Over 6000 Patients From Double-Blind and Open-Label Extension Studies. Circulation. 2017 May 9;135(19):1819-1831. doi: 10.1161/CIRCULATIONAHA.116.025233. Epub 2017 Mar 1. PMID 28249876
- [Background] Kasichayanula S, Grover A, Emery MG, Gibbs MA, Somaratne R, Wasserman SM, Gibbs JP. Clinical Pharmacokinetics and Pharmacodynamics of Evolocumab, a PCSK9 Inhibitor. Clin Pharmacokinet. 2018 Jul;57(7):769-779. doi: 10.1007/s40262-017-0620-7. PMID 29353350
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Japanese men or women ≥ 20 to ≤ 80 years of age and who were at high risk for cardiovascular events, on a stable dose of an approved statin (with or without ezetimibe) and fasting low-density lipoprotein cholesterol (LDL-C) ≥ 115 mg/dL.
  First patient enrolled on 10 July 2012; last patient enrolled 19 February 2013.
Pre-assignment Details: Randomization was stratified by screening LDL-C level (< 130 mg/dL [3.4 mmol/L] vs
  ≥ 130 mg/dL) and by diagnosis of heterozygous familial hypercholesterolemia (HeFH) (yes vs no).
Period: Overall Study
Arm/Group | Placebo Q2W | Placebo Q4W | Evolocumab 70 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 420 mg Q4W
Started | 52 | 51 | 50 | 52 | 52 | 53
Received Treatment | 52 | 50 | 49 | 52 | 51 | 53
Completed | 52 | 50 | 47 | 50 | 51 | 51
Not Completed | 0 | 1 | 3 | 2 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 3 | 1 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (all randomized participants who received at least 1 dose of investigational product).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Q2W | Placebo Q4W | Evolocumab 70 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 420 mg Q4W | Total
Number analyzed (Participants) | 52 | 50 | 49 | 52 | 51 | 53 | 307
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (10.1) | 60.9 (9.8) | 64.1 (9.7) | 60.8 (9.2) | 61.6 (9.6) | 61.3 (9.9) | 61.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 24 | 20 | 23 | 17 | 114
  Male | 36 | 36 | 25 | 32 | 28 | 36 | 193
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 52 | 50 | 49 | 52 | 51 | 53 | 307
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stratification Factor: LDL Level [Number; unit: participants]
  < 130 mg/dL | 17 | 17 | 15 | 17 | 15 | 17 | 98
  ≥ 130 mg/dL | 35 | 33 | 34 | 35 | 36 | 36 | 209
Stratification Factor: Diagnosis of Heterozygous Familial Hypercholesterolemia (HeFH) [Number; unit: participants]
  No | 48 | 47 | 47 | 49 | 47 | 49 | 287
  Yes | 4 | 3 | 2 | 3 | 4 | 4 | 20
LDL-C Concentration [Mean (Standard Deviation); unit: mg/dL] — LDL-C was measured using ultracentrifugation.
  mg/dL | 144.4 (18.1) | 141.8 (23.4) | 143.6 (20.6) | 140.7 (23.3) | 141.0 (21.2) | 139.7 (18.8) | 141.8 (20.9)
Non-High-Density Lipoprotein Cholesterol (non-HDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] | 171.3 (23.0) | 168.7 (26.1) | 170.6 (27.2) | 166.3 (26.2) | 165.5 (24.4) | 166.7 (23.5) | 168.2 (25.0)
Apolipoprotein B Concentration [Mean (Standard Deviation); unit: mg/dL] | 114.6 (15.4) | 112.5 (16.6) | 113.1 (19.2) | 109.4 (16.0) | 109.6 (16.9) | 109.8 (15.9) | 111.5 (16.7)
Very Low-Density Lipoprotein Cholesterol (VLDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] | 26.9 (10.5) | 27.1 (10.7) | 26.9 (13.3) | 25.6 (10.8) | 24.6 (10.5) | 27.0 (12.0) | 26.4 (11.3)
Total Cholesterol/HDL-C Ratio [Mean (Standard Deviation); unit: ratio] | 4.380 (0.949) | 4.317 (1.075) | 4.366 (1.177) | 4.302 (1.039) | 4.228 (0.993) | 4.210 (0.955) | 4.300 (1.026)
Apolipoprotein B/Apolipoprotein A-1 Ratio [Mean (Standard Deviation); unit: ratio] | 0.750 (0.150) | 0.741 (0.177) | 0.743 (0.177) | 0.722 (0.163) | 0.725 (0.151) | 0.714 (0.158) | 0.732 (0.162)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 12
Description: LDL-C was measured using ultracentrifugation.
Time Frame: Baseline and Week 12
Population: Full analysis set; missing ultracentrifugation (UC) LDL-C at Week 12 was imputed using last observation carried forward (LOCF) and calculated LDL-C.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo Q4W | Evolocumab 70 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 420 mg Q4W
Number analyzed (Participants) | 52 | 50 | 49 | 52 | 51 | 53
percent change | -2.71 (2.16) | 0.05 (2.32) | -55.56 (2.23) | -71.32 (2.16) | -58.10 (2.33) | -63.89 (2.27)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; The null hypothesis was that there was no mean difference in the percent change from Baseline at Week 12 in LDL-C between evolocumab and placebo, and the alternative hypothesis was that a mean difference did exist; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -68.61, 95% CI 2-sided [-74.51 to -62.71], Standard Error of Mean 2.99 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo Q2W vs Evolocumab 70 mg Q2W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -52.85, 95% CI 2-sided [-58.84 to -46.86], Standard Error of Mean 3.03 — Placebo is the reference
Statistical Analysis 3: Comparison: Placebo Q4W vs Evolocumab 420 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -63.94, 95% CI 2-sided [-70.23 to -57.66], Standard Error of Mean 3.18 — Placebo is the reference
Statistical Analysis 4: Comparison: Placebo Q4W vs Evolocumab 280 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -58.16, 95% CI 2-sided [-64.51 to -51.81], Standard Error of Mean 3.21 — Placebo is the reference

2. Secondary Outcome: Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 12
Description: LDL-C was measured using ultracentrifugation.
Time Frame: Baseline and Week 12
Population: Full analysis set; missing data were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo Q2W | Placebo Q4W | Evolocumab 70 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 420 mg Q4W
Number analyzed (Participants) | 52 | 50 | 49 | 52 | 51 | 53
mg/dL | -1.8 (3.6) | 0.8 (3.4) | -77.2 (3.7) | -98.0 (3.6) | -79.9 (3.4) | -87.4 (3.3)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -96.3, 95% CI 2-sided [-106.0 to -86.5], Standard Error of Mean 4.9 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo Q2W vs Evolocumab 70 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -75.5, 95% CI 2-sided [-85.4 to -65.5], Standard Error of Mean 5.0 — Placebo is the reference
Statistical Analysis 3: Comparison: Placebo Q4W vs Evolocumab 420 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -88.2, 95% CI 2-sided [-97.4 to -79.0], Standard Error of Mean 4.7 — Placebo is the reference
Statistical Analysis 4: Comparison: Placebo Q4W vs Evolocumab 280 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -80.7, 95% CI 2-sided [-90.0 to -71.4], Standard Error of Mean 4.7 — Placebo is the reference

3. Secondary Outcome: Percentage of Participants With an LDL-C Response at Week 12
Description: An LDL-C response was defined as LDL-C < 70 mg/dL (1.8 mmol/L) at Week 12. LDL-C was measured using ultracentrifugation.
Time Frame: Week 12
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Placebo Q4W | Evolocumab 70 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 420 mg Q4W
Number analyzed (Participants) | 52 | 50 | 49 | 52 | 51 | 53
percentage of participants | 0.0 (3.6) | 0.0 (3.4) | 66.0 (3.7) | 96.0 (3.6) | 80.4 (3.4) | 82.4 (3.3)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Testing based on a significance level of 0.05; Logistic Regression model includes treatment arms in dose frequency of Q2W and stratification factor of screening LDL-C level; Odds Ratio (OR) = 1945.68, 95% CI 2-sided [89.64 to 42232.63] — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo Q2W vs Evolocumab 70 mg Q2W; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Testing based on a significance level of 0.05; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 281.13, 95% CI 2-sided [14.74 to 5360.92] — Placebo is the reference
Statistical Analysis 3: Comparison: Placebo Q4W vs Evolocumab 420 mg Q4W; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Testing based on a significance level of 0.05; Logistic Regression model includes treatment arms in dose frequency of Q4W and stratification factor of screening LDL-C level; Odds Ratio (OR) = 536.45, 95% CI 2-sided [28.37 to 10143.40] — Placebo is the reference
Statistical Analysis 4: Comparison: Placebo Q4W vs Evolocumab 280 mg Q4W; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Testing based on a significance level of 0.05; [statistical method as in outcome 3, analysis 3]; Odds Ratio (OR) = 595.59, 95% CI 2-sided [31.11 to 11402.67] — Placebo is the reference

4. Secondary Outcome: Percent Change From Baseline to Week 12 in Non-HDL-C
Time Frame: Baseline and Week 12
Population: Full analysis set; missing data were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo Q4W | Evolocumab 70 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 420 mg Q4W
Number analyzed (Participants) | 52 | 50 | 49 | 52 | 51 | 53
percent change | -2.20 (1.94) | 0.55 (2.17) | -51.66 (2.00) | -64.76 (1.94) | -53.00 (2.17) | -57.53 (2.12)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -62.56, 95% CI 2-sided [-67.85 to -57.27], Standard Error of Mean 2.68 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo Q2W vs Evolocumab 70 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -49.46, 95% CI 2-sided [-54.83 to -44.08], Standard Error of Mean 2.72 — Placebo is the reference
Statistical Analysis 3: Comparison: Placebo Q4W vs Evolocumab 420 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -58.08, 95% CI 2-sided [-63.93 to -52.22], Standard Error of Mean 2.96 — Placebo is the reference
Statistical Analysis 4: Comparison: Placebo Q4W vs Evolocumab 280 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -53.54, 95% CI 2-sided [-59.46 to -47.63], Standard Error of Mean 2.99 — Placebo is the reference

5. Secondary Outcome: Percent Change From Baseline to Week 12 in Apolipoprotein B
Time Frame: Baseline and Week 12
Population: Full analysis set; missing data were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo Q4W | Evolocumab 70 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 420 mg Q4W
Number analyzed (Participants) | 52 | 50 | 49 | 52 | 51 | 53
percent change | -0.90 (1.82) | 0.22 (2.02) | -47.65 (1.88) | -61.59 (1.82) | -47.16 (2.03) | -53.22 (1.98)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -60.69, 95% CI 2-sided [-65.67 to -55.72], Standard Error of Mean 2.52 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo Q2W vs Evolocumab 70 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -46.75, 95% CI 2-sided [-51.80 to -41.70], Standard Error of Mean 2.56 — Placebo is the reference
Statistical Analysis 3: Comparison: Placebo Q4W vs Evolocumab 420 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -53.44, 95% CI 2-sided [-58.91 to -47.97], Standard Error of Mean 2.77 — Placebo is the reference
Statistical Analysis 4: Comparison: Placebo Q4W vs Evolocumab 280 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -47.37, 95% CI 2-sided [-52.90 to -41.85], Standard Error of Mean 2.80 — Placebo is the reference

6. Secondary Outcome: Percent Change From Baseline to Week 12 in VLDL-C
Time Frame: Baseline and Week 12
Population: Full analysis set; missing data were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo Q4W | Evolocumab 70 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 420 mg Q4W
Number analyzed (Participants) | 52 | 50 | 49 | 52 | 51 | 53
percent change | 8.23 (8.55) | 7.26 (6.87) | -16.02 (8.74) | -26.26 (8.44) | -13.56 (6.80) | -22.56 (6.71)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority or Other; p = 0.004, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -34.49, 95% CI 2-sided [-57.71 to -11.26], Standard Error of Mean 11.75 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo Q2W vs Evolocumab 70 mg Q2W; Test type: Superiority or Other; p = 0.044, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -24.25, 95% CI 2-sided [-47.83 to -0.68], Standard Error of Mean 11.93 — Placebo is the reference
Statistical Analysis 3: Comparison: Placebo Q4W vs Evolocumab 420 mg Q4W; Test type: Superiority or Other; p = 0.002, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -29.82, 95% CI 2-sided [-48.32 to -11.32], Standard Error of Mean 9.36 — Placebo is the reference
Statistical Analysis 4: Comparison: Placebo Q4W vs Evolocumab 280 mg Q4W; Test type: Superiority or Other; p = 0.028, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -20.82, 95% CI 2-sided [-39.41 to -2.22], Standard Error of Mean 9.41 — Placebo is the reference

7. Secondary Outcome: Percent Change From Baseline to Week 12 in Total Cholesterol/HDL-C Ratio
Time Frame: Baseline and Week 12
Population: Full analysis set; missing data were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo Q4W | Evolocumab 70 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 420 mg Q4W
Number analyzed (Participants) | 52 | 50 | 49 | 52 | 51 | 53
percent change | -4.82 (1.91) | 1.19 (2.09) | -42.04 (1.98) | -51.81 (1.91) | -44.11 (2.10) | -45.47 (2.05)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -46.98, 95% CI 2-sided [-52.21 to -41.76], Standard Error of Mean 2.64 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo Q2W vs Evolocumab 70 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -37.22, 95% CI 2-sided [-42.52 to -31.91], Standard Error of Mean 2.68 — Placebo is the reference
Statistical Analysis 3: Comparison: Placebo Q4W vs Evolocumab 420 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -46.66, 95% CI 2-sided [-52.32 to -41.00], Standard Error of Mean 2.86 — Placebo is the reference
Statistical Analysis 4: Comparison: Placebo Q4W vs Evolocumab 280 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -45.30, 95% CI 2-sided [-51.02 to -39.58], Standard Error of Mean 2.89 — Placebo is the reference

8. Secondary Outcome: Percent Change From Baseline to Week 12 in Apolipoprotein B/Apolipoprotein A-1 Ratio
Time Frame: Baseline and Week 12
Population: Full analysis set; missing data were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo Q4W | Evolocumab 70 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 420 mg Q4W
Number analyzed (Participants) | 52 | 50 | 49 | 52 | 51 | 53
percent change | -3.18 (2.12) | 1.44 (2.21) | -50.71 (2.19) | -64.53 (2.12) | -50.79 (2.22) | -56.31 (2.16)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -61.35, 95% CI 2-sided [-67.14 to -55.56], Standard Error of Mean 2.93 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo Q2W vs Evolocumab 70 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -47.53, 95% CI 2-sided [-53.41 to -41.65], Standard Error of Mean 2.98 — Placebo is the reference
Statistical Analysis 3: Comparison: Placebo Q4W vs Evolocumab 420 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -57.75, 95% CI 2-sided [-63.73 to -51.77], Standard Error of Mean 3.03 — Placebo is the reference
Statistical Analysis 4: Comparison: Placebo Q4W vs Evolocumab 280 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factor of screening LDL-C level; LS Mean Treatment Difference = -52.22, 95% CI 2-sided [-58.27 to -46.18], Standard Error of Mean 3.06 — Placebo is the reference

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Evolocumab Q2W 70 MG: Participants received 70 mg evolocumab by subcutaneous injection once every 2 weeks for 12 weeks.
- Evolocumab Q2W 140 MG: Participants received 140 mg evolocumab by subcutaneous injection once every 2 weeks for 12 weeks.
- Evolocumab Q4W 280 MG: Participants received 280 mg evolocumab by subcutaneous injection once every 4 weeks for 12 weeks.
- Evolocumab Q4W 420 MG: Participants received 420 mg evolocumab by subcutaneous injection once every 4 weeks for 12 weeks.
Arm/Group | Placebo Q2W | Placebo Q4W | Evolocumab Q2W 70 MG | Evolocumab Q2W 140 MG | Evolocumab Q4W 280 MG | Evolocumab Q4W 420 MG
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/50 | 0/49 | 1/52 | 1/51 | 2/53
Other Adverse Events (participants affected / at risk) | 6/52 | 6/50 | 10/49 | 9/52 | 12/51 | 8/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=52) | Placebo Q4W (N=50) | Evolocumab Q2W 70 MG (N=49) | Evolocumab Q2W 140 MG (N=52) | Evolocumab Q4W 280 MG (N=51) | Evolocumab Q4W 420 MG (N=53)
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Carcinoid tumour of the caecum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=52) | Placebo Q4W (N=50) | Evolocumab Q2W 70 MG (N=49) | Evolocumab Q2W 140 MG (N=52) | Evolocumab Q4W 280 MG (N=51) | Evolocumab Q4W 420 MG (N=53)
Nasopharyngitis (Infections and infestations) | 6 | 6 | 10 | 9 | 12 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.